CLINICAL TRIAL: NCT03718598
Title: Effectiveness of Home Exercise in Pregnant Women With Carpal Tunnel Syndrome
Brief Title: Carpal Tunnel Syndrome in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 9671
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Carpal Tunnel Syndrome; Exercise
Keywords: Carpal tunnel syndrome; home exercise; pregnant women
MeSH Terms: conditions — Carpal Tunnel Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carpal tunnel syndrome: Patients with mild and moderate carpal tunnel syndrome
  Interventions: Behavioral: Tendon and Nerve Gliding Exercises
- normal: Patients without mild and moderate carpal tunnel syndrome
  Interventions: Behavioral: Tendon and Nerve Gliding Exercises

INTERVENTIONS:
Behavioral: Tendon and Nerve Gliding Exercises — Tendon and Nerve Gliding Exercises: The tendon slip exercises used in this study were performed in five different positions, namely flexion, flat, hook, punch, table top and flat punch positions. Nerve-gliding exercises were performed by moving the fingers and wrists in six different positions, focusing on the median nerve consisting of all the disease grip, finger lengthening, wrist extension, thumb extension, forearm supination and gentle gentle gait. Instructions were given to make 10 sets of exercises in 3 sets, written and verbal, in order to have e exercises for all patient's tendons and nerves shifting exercises. Brochures were also provided explaining the exercises.

SUMMARY:
The purpose of our study is to evaluate the effectiveness of the home exercise program in patients who develop Carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
Materials and Method: Thirty-three patients with CTS (mild to moderate) were included to randomized, single-blind, controlled clinical trial. Based on EMG results and clinical examination, patient group was divided two part as mild and moderate CTS (group 1) and normal (group 2). The Sick Boston Carpal Tunnel Syndrome Questionnaire form was filled in face-to-face method.

Cases in this study: Patients who had pain and numbness problems at the hands of the Bezmiâlem Vakif University Polyclinic for Women and Obstetrics were then directed to the Bezmiâlem Vakif University Physical Therapy Rehabilitation Policlinic. After the examination and clinical testing of each patient (Tinel test, Phalen's test, Reverse Phalen's and Durkan's Carpal Compression test), the patients were directed to Bezmiâlem Vakif University Neurology Policlinic. Based on electromyography (EMG) results and clinical examination, the group was classified as mild and moderate CTS (group 1) and normal (group 2). A disease exercise form was distributed for all patients to do exercises.

ELIGIBILITY:
Inclusion Criteria:

* Provocation tests during the examination and physical examination to match the median nerve distribution those who have symptoms of numbness, tingling, weakness and pain in the hands that have lasted at least 1 month.
* Patients with confirmed mild-moderate idiopathic CTS on EMG.

Exclusion Criteria:

* Previously undergone carpal tunnel surgery
* Gestational diabetes mellitus,
* Eclampsia, preeclampsia
* Thyroid disorders
* Arthropathies
* Hand or wrist trauma
* Bilateral fractures
* Severe cts
* Atrial fibrillation
* Cervical radiculopathy
* Peripheral neuropathy
* Thoracic outlet syndrome
* Diabetes mellitus
* Hypothyroidism
* Hyperthyroidism
* Rheumatologic disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Non-Probability Sample: Any of a variety of other sampling processes, such as convenience sampling or invitation to volunteer
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Sick Boston Carpal Tunnel Syndrome Questionnaire | Patients were evaluated before treatment and 1 month after the birth.
  It is a test consisting of two parts evaluating symptom severity (BSSS) and functional capacity (BFCS). BSSS consists of 11 questions for symptoms. In each question there are five different answers with scores between 1 and 5. The average score is obtained by dividing the total score by the number of questions. High score indicates severe symptom. BFCS consists of 8 questions for functional capacity. Again, there are five different answers in each question, ranging from 1 to 5. The average score is obtained by dividing the total score by the number of questions. The high score indicates that the functional capacity decreases. The questionnaire has been validated and tested for Turkish society (15). The questionnaire has been validated and tested for Turkish society (16).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR